CLINICAL TRIAL: NCT02262455
Title: An Open-Label Multiple Ascending Dose Phase 1/1B Pharmacokinetic and Pharmacodynamic Study of STM 434, an Activin Type 2B Receptor Fc Fusion, Alone and in Combination With Liposomal Doxorubicin in Patients With Ovarian Cancer or Other Advanced Solid Tumors
Brief Title: Effects of STM 434 Alone or in Combination With Liposomal Doxorubicin in Patients With Ovarian Cancer or Other Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santa Maria Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STM-434-001
Record Dates: First submitted 2014-09-29; First posted 2014-10-13 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Endometrial Cancer; Solid Tumors
Keywords: Serous tumor; Granulosa tumor; Clear Cell tumor; Endometrial cancer; Advanced solid tumors; Adenocarcinoma; Prostate cancer; Head and Neck cancer; Lung cancer; Non-small cell lung cancer; Small cell lung cancer; Gastric cancer; Kidney cancer; Pancreatic cancer; Breast cancer; Colorectal cancer; Bladder cancer; Esophagus cancer; Liver cancer; Hepatobiliary cancer; Skin cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms; Adenocarcinoma; Prostatic Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Stomach Neoplasms; Kidney Neoplasms; Pancreatic Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Urinary Bladder Neoplasms; Esophageal Neoplasms; Liver Neoplasms; Skin Neoplasms | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- STM 434 (Experimental)
  Interventions: Drug: STM 434
- STM 434 and Liposomal Doxorubicin (Experimental)
  Interventions: Drug: STM 434; Drug: Liposomal doxorubicin

INTERVENTIONS:
Drug: STM 434 — STM 434 will be administered by IV injection. There are five planned dose levels, from 0.25mg/kg to 4mg/kg, which is dependent on the cohort (group) a participant is assigned to.
Drug: Liposomal doxorubicin — Liposomal doxorubicin (40 mg/m2) will be administered once every 28 days by IV infusion prior to STM 434 for those participants enrolled in Part 3 of the trial. Liposomal doxorubicin will be administered for a maximum of 6 cycles (each cycle being 28 days).
  Arms: STM 434 and Liposomal Doxorubicin

SUMMARY:
This is a Phase I study to test the safety, pharmacokinetics and effectiveness of STM 434 alone, or in combination with liposomal doxorubicin, in patients with ovarian cancer or other advanced solid tumors.

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known) study to evaluate the safety, pharmacokinetics (study of what the body does to a drug), pharmacodynamics (study of what a drug does to the body), and anti-tumor activities of STM 434 (an inhibitor of activin A) in patients with ovarian cancer and other advanced solid tumors. The study will be conducted in 3 phases (Part 1, Part 2 and Part 3). In the first part of the study (Part 1), which will enroll patients with multiple solid tumor types, the maximum tolerated dose (MTD) of STM 434 will be determined for use in the second and third parts of the study (Parts 2 and 3). In the second part (Part 2), which will enroll patients with ovarian cancer, STM 434 will be administered alone, and in the third part (Part 3), which will enroll patients with ovarian cancer, STM 434 will be given together with a chemotherapy called liposomal doxorubicin. Doses of STM 434 (starting at 0.25 mg/kg up to a maximum of 4 mg/kg) will be taken on one of three dosing schedules to determine the MTD. Patients will continue taking STM 434 until their tumor progresses. Serial blood samples will be collected for pharmacokinetic and pharmacodynamic testing and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Males and postmenopausal females, 18 years or older
* Advanced solid tumors with histologic diagnosis confirming cancer
* Patients with recurrent metastatic or locally advanced disease considered refractory or intolerant to all standard treatment available for their tumor, or those tumors for which no standard treatment is available
* Subjects with serous ovarian/fallopian tube/primary peritoneal, granulosa cell tumors or clear cell tumors considered platinum refractory/resistant, defined as having at least one prior platinum-based chemotherapeutic regimen with a subsequent platinum-free interval of < 12 months, having progression during platinum-based therapy, or having persistent disease after a platinum-based therapy, are eligible. Intolerant subjects, defined as unable to receive further platinum due to toxicity, are eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Informed consent

Exclusion Criteria:

* History of gastrointestinal bleeding within the past 6 months
* History of epistaxis requiring medical/surgical intervention (such as nasal packing) within the past 6 months
* History of central nervous system hemorrhage
* History of bleeding diathesis or known qualitative platelet defect (including von Willebrand disease)
* Ongoing need for therapeutic anticoagulants (full dose heparin, warfarin, factor Xa or direct thrombin inhibitors; rivaroxaban, apixaban, dabigatran) chronic use of aspirin or anti-platelet agents (ticlopidine or clopidogrel)
* History of hereditary hemorrhagic telangiectasia (HHT, Osler-Weber-Rendu syndrome)
* Myocardial infarction, unstable angina within the past 6 months, or congestive heart failure New York Heart Association Class II or greater
* Chemotherapy, hormonal therapy or radiation therapy within the past 3 weeks, antibody/biologic therapy within 5 half-lives or within the past 4 weeks (whichever is longer)
* Current bowel obstruction
* Brain metastasis
* Known HIV infection and/or active Hepatitis B or C infection
* Prior treatment with any investigational product within the past 4 weeks
* Not willing to use contraception (inclusive of abstinence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-01-13 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | MTD will be assessed for STM 434 alone in Part 1 and in combination with liposomal doxorubicin in Part 3 once the last subject in each cohort completes 28 days of treatment.
  To define the maximum tolerated dose (MTD) of STM 434 administered alone or in combination with liposomal doxorubicin chemotherapy in patients with ovarian cancer or other advanced solid tumors.

SECONDARY OUTCOMES:
Recommended Phase 2 dose (RP2D) | RP2D will be assessed in Part 1 once the last subject in each cohort completes 28 days of treatment.
  To define the recommended Phase 2 dose (RP2D) in the event that there is no maximum tolerated dose (MTD) reached.
Radiographic response rate | Efficacy parameters will be assessed at three points in the study: once Part 1 and Part 3 are fully enrolled, and during Part 2 of the study. On average the review is expected to occur once every 8 months, for up to 24 months.
  To collect preliminary radiographic response data, including CT, MRI scans, during therapy with STM 434.
Muscle function and body composition | Efficacy parameters will be assessed at three points in the study: once Part 1 and Part 3 are fully enrolled, and during Part 2 of the study. On average the review is expected to occur once every 8 months for up to 24 months.
  To collect preliminary anti-cachexia data, including body composition and laboratory parameters, during therapy with STM 434.

CONTACTS AND LOCATIONS:
Overall Officials: Willis Navarro, MD, Study Director — Santa Maria Biotherapeutics
Locations (4):
- United States (4):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

REFERENCES:
- [Derived] Bian X, Snow ZK, Zinn CJ, Gowan CC, Conley SM, Bratulin AL, Elhusseiny KM, Miller J, Tchkonia T, Kirkland JL, Lerman LO, Hickson LJ. Activin A Antagonism with Follistatin Reduces Kidney Fibrosis, Injury, and Cellular Senescence-Associated Inflammation in Murine Diabetic Kidney Disease. Kidney360. 2025 Mar 28;6(8):1278-1291. doi: 10.34067/KID.0000000776. PMID 40152935
- [Derived] Tao JJ, Cangemi NA, Makker V, Cadoo KA, Liu JF, Rasco DW, Navarro WH, Haqq CM, Hyman DM. First-in-Human Phase I Study of the Activin A Inhibitor, STM 434, in Patients with Granulosa Cell Ovarian Cancer and Other Advanced Solid Tumors. Clin Cancer Res. 2019 Sep 15;25(18):5458-5465. doi: 10.1158/1078-0432.CCR-19-1065. Epub 2019 May 8. PMID 31068369